CLINICAL TRIAL: NCT01887509
Title: Evaluation of Rectal Tumor Margin Using Confocal Endomicroscopy and Comparison to Histopathology
Acronym: TRaMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with patients recruitment, study acceptance and protocol implementation.
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-005; 2013-A00406-39 (Other: ANSM France)
Record Dates: First submitted 2013-06-20; First posted 2013-06-27 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Rectal Cancer; Rectal Adenocarcinoma
Keywords: Rectal cancer; Tumor margin; Confocal endomicroscopy; Virtual biopsy; Fluorescein
MeSH Terms: conditions — Rectal Neoplasms | interventions — Proctoscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Probe-based confocal laser endomicroscopy — Patients will undergo:
  * Conventional rectoscopy
  * pCLE exam following injection of fluorescein, fluorescent contrast agent
  * EUS : echoendoscopy
  * Biopsies for histopathology : location identical to those of pCLE
  * Tumor resection will be performed according to standard oncologic principles.
  All visible lesions will be documented. Both healthy and tumor tissue will be examined. Location of sites of interest will be documented on a schema, completed with photographs of endoscopic view.
  Biopsies will be harvested in both healthy and tumor tissue as well.
  After all procedures are complete, a second assessment of pCLE images by a third party will be performed.
  Other Names: Cellvizio® with ColoFlex probe
Procedure: Rectoscopy — Patients will undergo:
  * Conventional rectoscopy
  * pCLE exam following injection of fluorescein, fluorescent contrast agent
  * EUS : echoendoscopy
  * Biopsies for histopathology : location identical to those of pCLE - Tumor resection will be performed according to standard oncologic principles.
  All visible lesions will be documented. Both healthy and tumor tissue will be examined. Location of sites of interest will be documented on a schema, completed with photographs of endoscopic view.
  Both healthy and tumor tissue will be examined.
Procedure: EUS — Patients will undergo:
  * Conventional rectoscopy
  * pCLE exam following injection of fluorescein, fluorescent contrast agent
  * EUS : echoendoscopy
  * Biopsies for histopathology : location identical to those of pCLE - Tumor resection will be performed according to standard oncologic principles.
  All visible lesions will be documented. Both healthy and tumor tissue will be examined. Location of sites of interest will be documented on a schema, completed with photographs of endoscopic view.
  Other Names: Echoendoscopy
Procedure: Biopsy and resection — Patients will undergo:
  * Conventional rectoscopy
  * pCLE exam following injection of fluorescein, fluorescent contrast agent
  * EUS : echoendoscopy
  * Biopsies for histopathology : location identical to those of pCLE
  * Tumor resection will be performed according to standard oncologic principles.
  All visible lesions will be documented. Both healthy and tumor tissue will be examined. Location of sites of interest will be documented on a schema, completed with photographs of endoscopic view.
  Biopsies will be harvested in both healthy and tumor tissue as well.

SUMMARY:
This innovative study will involve the use of probe-based confocal laser endomicroscopy, a new medical imaging technology never used for surgical indications to date. Virtual biopsies (pCLE images) will be compared to histopathology analysis.

This study focuses on the evaluation of rectal tumor margins. The hypothesis is that pCLE will allow identification of rectal tumor margin, comparable to that of histopathology. In the future, decision of resection margin could rely on intraoperative pCLE exam.

The proposed study is a feasibility study, first in the indication of rectal cancer.

DETAILED DESCRIPTION:
Defining the limits of resection of rectal tumors is often imprecise. The identification of the banks of a tumor becomes critical when it comes to the decision to potentially sacrifice the sphincter during the surgical resection. Currently tumor margins are identified by direct examination by the surgeon, or using flexible endoscopy. Endoscopy and confocal microscopy could provide precise images of tumor enabling the reliable definition of resection margins.

There would be a direct benefit for the patient, whom sphincter could be preserved. pCLE (probe-based Confocal Laser Endomicroscopy) has already been widely used for colorectal lesions, and its value proposition has been demonstrated and validated in several studies. This study is the first using pCLE intraoperatively. Study results may lead the use of pCLE to validate surgical procedure decision (resection margin) and to a revision of patient management for colorectal cancer, by adapting neoadjuvant radiochemotherapy to the patient's responder status.

The goal is to identify tumor margin (lower pole) to optimize the resection margin, and to limit resection of healthy rectal tissue for optimal anal sphincter preservation. Moreover, determining the optimal date of surgery following neoadjuvant radiochemotherapy in rectal cancer is being discussed and no consensus has been reached. Therefore, to date, there is no formal evaluation of tumor response. This is partly due to the lack of information on tumor state and tumor evolution over time, between the end of radiochemotherapy and surgery. Histological follow up of tumor would provide supporting information to fill this gap. However, frequent tumor biopsies are not possible. Alternatively, probe-based confocal laser endomicroscopy (pCLE) could allow for a sequential analysis of tumor response. Response to treatment could be assessed and used to define optimal date of surgical resection, depending on patient responding status to treatment. Responding patients would undergo surgery at a later date than non-responders, in whom surgery could be performed earlier.

Benefits of the study lay in the more accurate definition of resection margins, with its associated potential therapeutic impact of the anal sphincter preservation and in the definition of the optimal date of rectal tumor resection, based on response status to radiochemotherapy.

Study interests are :

* Microscopic structure of tumor will be analyzed at the cellular and microvascular levels and compared to healthy mucosa.
* Evolution of response during and following radiochemotherapy will be assessed, and will help classify patients as responders/non responders.
* pCLE results will be compared to histopathology results on pre-treatment and resection biopsies.
* Images gathered through the imaging modalities (WLE, pCLE, EUS) along with histopathology results will be combined to create an atlas and database of rectal tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female over 18 years old
* Patient with rectal adenocarcinoma :

  * stage T1 or T2, N0 (one single evaluation, during resection)
  * stage N+ or T3 (pre- and post-radiochemotherapy evaluations)
* Absence of contra-indication to rectoscopy conduct
* Patient able to understand the study and to provide written informed consent
* Patient registered with the French social security regime

Non-inclusion criteria:

* Absence of written informed consent
* Patient with known or suspected allergy to fluorescein
* Patient with history of reaction jeopardizing the vital prognosis during angiography
* Patient with history of multiple or serious allergic reaction to drugs
* Patient presenting, in the investigator's judgment, a condition or disease preventing their participation to study procedures
* Patient pregnant or breast-feeding
* Patient within exclusion period from other clinical trial
* Patient having forfeited their freedom of an administrative or legal obligation
* Patient being under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-11-07 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Concordance in identification of lower pole of tumor | Up to 9 months
  Identification of lower pole of tumor will be compared between pCLE (optical images, virtual biopsies) and conventional histopathology (biopsies, postoperative analysis of resected piece). Samples of tumor tissue and closest tissue thought to be disease-free.
  Conventional biopsies and virtual biopsies prior to radiochemotherapy start (if applicable) and during surgery.

SECONDARY OUTCOMES:
Identification of tissue characteristics | Up to 9 months
  Microvascularisation density, general microstructure, image interpretation criteria, true/false positive/negative.
  Will be assessed for all patients at the time of surgical procedure. Also prior to treatment for patients undergoing radiochemotherapy.
Concordance of techniques (pCLE and histopathology) | Up to 9 months
  Evaluation of concordance between pCLE and conventional histopathology for :
  * tissue characterization prior to and after radiochemotherapy, if applicable
  * radiochemotherapy response assessment
  * resection margin evaluation
  For patients undergoing radiochemotherapy, 2 exams: prior to treatment start and during surgery For patients with surgery only, 1 exam: during surgery
Comparison of pCLE results to EUS (echoendoscopy) results | Upon surgery
  pCLE results will be compared to EUS prior to radiochemotherapy and at the time of resection.
Creation of an image bank | Up to 9 months
  Creation of an image bank : identification of quality and safety criteria to be of interest for use at the time of resection
Assessment of predictive value of interpretation criteria | Up to 9 months
  Results will be analyzed to assess whether pCLE interpretation criteria have a predictive value for identification of responder/non-responders patients to radiochemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Joël Leroy, Pr, Principal Investigator — Service de Chirurgie Disgestive et Endocrinienne - Nouvel Hôpital Civil - Strasbourg
Locations (1):
- Service de chirurgie digestive et endocrinienne - Nouvel Hôpital Civil, Strasbourg, France

REFERENCES:
- [Result] Wijsmuller AR, Ghnassia JP, Varatharajah S, Schaeffer M, Leroy J, Marescaux J, Ignat M, Mutter D. Prospective Trial on Probe-Based Confocal Laser Endomicroscopy for the Identification of the Distal Limit in Rectal Adenocarcinoma. Surg Innov. 2018 Aug;25(4):313-322. doi: 10.1177/1553350618773011. Epub 2018 May 7. PMID 29732957